CLINICAL TRIAL: NCT01844336
Title: PBASE System Idiopathic Rhinitis Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR003
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Idiopathic Rhinitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBASE system 1.1 + CT100 (active treatment) (Experimental)
  Interventions: Device: PBASE system 1.1 + CT100 (active treatment)
- PBASE system 1.1 + CT100 (placebo treatment) (Placebo Comparator)
  Interventions: Device: PBASE system 1.1 + CT100 (placebo treatment)

INTERVENTIONS:
Device: PBASE system 1.1 + CT100 (active treatment)
  Arms: PBASE system 1.1 + CT100 (active treatment)
Device: PBASE system 1.1 + CT100 (placebo treatment)
  Arms: PBASE system 1.1 + CT100 (placebo treatment)

SUMMARY:
The purpose of this study is to evaluate the performance of the PBASE system, in terms of the efficacy of treatment in patients with idiopathic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent (>12w) symptoms of idiopathic rhinitis dominated by nasal congestion (± secretion) for an average of at least 1 h per day for at least 5 days during a period of 14 days
* Having nasal congestion as major symptom, and a nasal congestion score of at least 2 (scale 0-3)
* Male or female 18 - 65 years
* Judged by the Investigator as suitable for participation in the study without safety concerns based on medical history and physical examination.
* Willing and able to provide written informed consent prior to participation in the clinical investigation
* Willing and able to comply with all study related procedures

Exclusion Criteria:

* Patients with Allergic rhinitis, demonstrated by either positive skin prick test, phadiatop or RAST
* Ongoing respiratory tract infection including nasal cavity at inclusion (treatment visit 1)
* Systemic steroid treatment less than 4 weeks before the inclusion in the study
* Patients with a history of nasal surgery like: septoplasty, cosmetic surgery, conchal surgery or any other nasal surgery except closed reposition for nasal fracture
* History of frequent nose bleeds or a condition that increases the risk of excessive bleeding
* Pronounced anterior septal deviation or other significant nasal pathology at endoscopic examination
* Current malignancy of any kind
* Known allergy to polyvinylchloride or medicinal liquid paraffin
* Any disease, condition (medical or surgical) which, in the opinion of the investigator, might compromise the study results, or would place the subject at increased risk.
* Any implant with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulation, spinal stimulator, bone growth stimulator, or cochlear implant or any other implant in the head-, and neck region.
* Previous treated with radiation on the face, head or neck regions
* Female patients who are pregnant or nursing, or become pregnant at any time from inclusion of the study until end of the 8 week follow-up visit
* Female patients: unwilling to use adequate contraceptive from the signing of the informed consent until end of the 8 week follow-up visit
* Received study drug in a clinical trial for an investigational drug within the previous 30 days, or 5 half-lives, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in total vasomotor rhinitis symptom score to visit 3 | From baseline to 28 days after treatment visit 1

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Falun
  - Gothenburg
  - Lund
  - Stockholm
  - Västerås